CLINICAL TRIAL: NCT02233855
Title: NACC 002: A Multicenter Prospective Natural History Study of Patients Presenting With Neurocysticercosis in North America
Brief Title: People Presenting With Neurocysticercosis in North America
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140191; 14-I-0191
Record Dates: First submitted 2014-09-06; First posted 2014-09-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-06-13

CONDITIONS: Neurocysticercosis
Keywords: Seizures; Cestode; Hydrocephalus; Taenia Solium; Helminth
MeSH Terms: conditions — Neurocysticercosis; Seizures; Cestode Infections; Hydrocephalus; Taeniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Neurocysticercosis (NCC) is caused by tapeworms that infect people. NCC can lead to serious brain problems such as seizures, sevre headaches and difficulties with movements or sensation in the limbs. Researchers want to learn more about the different ways in which people in the United States present with this disease and how they respond to standard and newer treatments.

Objective:

- To learn about the different forms of NCC that occurs throughout North America and how patients with these forms respond to treatment.

Eligibility:

- Adults age 18 or older with NCC.

Design:

* Participants will be screened with:
* Medical history and physical exam.
* A computed tomography (CT) brain scan The participant will lie still on a table that slides into a large donut-shaped scanner.
* Blood drawn through an arm vein for analysis
* A magnetic resonance imaging (MRI) scan of the brain and spine. They will lay flat in a long metal cylinder as the machine makes images of the body. During the scan, participants will receive a contrast agent through an IV that allows high resolution imaging of the brain and spine
* Participants will visit the clinic at 0, 1, 2, 3, 6, 12, and 24 months (7 times), and depending on the need for monitoring, more times. Participants will receive a schedule that will explain the procedures done at each visit.
* At these visits, participants may:
* Repeat the screening procedures.
* Be asked about their NCC symptoms and their physical and mental health.
* Have a urine test.
* Take a test of their ability to concentrate, their memory and spatial recognition.
* Have a lumbar puncture, if indicated by the state and severity of infection. A needle will be inserted through the skin and into the space between the bones in the back. Cerebrospinal fluid will be removed.

DETAILED DESCRIPTION:
Neurocysticercosis (NCC) is the most common helminthic CNS infection and the main cause of adult-onset seizures in low-to-middle income countries. Studies have documented significant endemicity in Latin America, Eastern Europe, sub-Saharan Africa, India and other parts of the world. The prevalence of NCC in North America is rising as a result of increased migration of people with the disease and, occasionally, immigration of individuals with asymptomatic tapeworms. Despite the gains in knowledge and understanding of the epidemiology, pathophysiology, diagnosis, and treatment, clinical care continues to be hampered by unanswered fundamental questions related to optimal diagnosis, staging, treatment, and follow-up of patients with NCC.

This multi-center, natural history study seeks to characterize: the frequency of the various forms of NCC in North American populations; the spectrum of treatment and management strategies across the North American Cysticercosis Consortium; and the response to therapy by evaluating a number of endpoints related to disease evolution and treatment, such as burden of disease, cognitive changes, radiographic changes, and treatment complications. This study will inform future research studies needed to eventually establish standardized management protocols for each form of this complex infection.

Subjects will have visits at screening, baseline, 1, 2 (optional), 3, 6, 12, and 24 months. Evaluations will include assessment of clinical status, antigen assays, radiographic imaging, functional assessments, immunologic evaluations, cognitive assessments, and quality of life measures. Additional clinically indicated visits may be scheduled as needed. This study does not provide any interventional therapies but will collect data on the course of treatment. Diagnostic examinations, consultations and medical treatment will be determined by the study clinician. Any samples removed for medical indications related to NCC may be evaluated for research purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults greater than or equal to18 years of age.
  2. Subject, or Subject s Legally Authorized Representative (LAR)/ Durable Power of Attorney (DPA), is able to provide informed consent and agree to allow samples to be stored for future research.
  3. Previously or currently diagnosed with definitive or probable NCC by a practitioner at NACC in accordance with the Del Brutto criteria modified for use in a North American populations.

For the purpose of this study, definitive and probable diagnostic certainty based on presence of criteria below.

Definitive diagnosis

1. Presence of 1 absolute criterion
2. Presence of 2 major + 1 minor + 1 epidemiological criterion

Probable diagnosis Presence of 1 major + 2 minor criterion

1. Presence of 1 major + 1 minor + 1 epidemiological criterion
2. Presence of characteristic calcification(s)

Del Brutto Diagnostic criteria

1. Absolute criteria

   1. Biopsy of a brain or spinal cord lesion
   2. Cystic lesion with scolex on CT or MRI
   3. Fundoscopic examination (subretinal parasites)
2. Major criteria

   1. Highly suggestive lesions on neuroimaging
   2. Positive serum enzyme-linked immunotransfer blot (EITB) assay
   3. Resolution of intracranial cysts after therapy
   4. Spontaneous resolution of small single enhancing lesions
3. Minor criteria

   1. Compatible lesions on neuroimaging
   2. Clinical manifestations suggestive for NCC (eg, headaches, seizures, neurological symptoms)
   3. Positive CSF ELISA for specific Ag/Ab
   4. Cysts outside CNS
4. Epidemiological criteria

   1. Evidence of household contact with T. solium
   2. Individuals coming from/living in endemic areas
   3. History of frequent travel to endemic areas
5. Single or multiple characteristic calcifications in subjects who meet epidemiologic criteria (4) without another identifiable etiology will be considered NCC in the case of calcified granulomas

EXCLUSION CRITERIA:

1. Subjects that in the opinion of the investigator have contraindications for participation in the study will be excluded, such as patients with current substance abuse or patients currently undergoing cancer chemotherapy.

Justification for Exclusion or Inclusion of Special Populations

Children

Children are eligible to participate in this clinical trial but will not be enrolled at the NIH because the NIH investigators do not see nor specialize in pediatric populations. In addition, NCC in the U.S. generally afflicts travelers and immigrants and is therefore exceedingly rare in pediatric populations in the U.S.

Adults Unable To Provide Consent-

Patients will be offered standard of care treatment delivered irrespective of cognitive status, including lumbar punctures that are used clinical management decisions as determined by the site PI. Exclusion of patients unable to provide consent because of cognitive impairment would limit the study population significantly, and potentially compromise the generalizability of results from this observational study. In cases where cognitive function precludes informed consent we will seek consent from the designated legal guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09-03; Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
The heterogeneity and complexity of the different forms of NCC will make it necessary to use different endpoints in analyzing the data collected from patients with each subtype of NCC. The endpoints listed here will be tailored and applied to th... | Throughout the course of the study

SECONDARY OUTCOMES:
To characterize the spectrum of diagnostic and treatment approaches across sites, including type and length of anthelmintic, anti-inflammatories, and anticonvulsants | Throughout the course of the study.
To determine exposure risks and estimate time to clinical symptomatic disease (incubation time) for each form of NCC | Throughout the course of the study.
For each form of NCC, to assess patient outcomes relative to: a) duration and type of anthelmintic therapy; b) duration and type of immunosuppressive therapy; and c) anticonvulsant therapy | Throughout the course of the study.
To correlate clinical features with radiographic findings at presentation, during treatment and follow-up for each form of NCC | Throughout the course of the study.
Determine proportion of patients with clinical and radiographic success 1 and 2 years after initiation of therapy. Definition of radiographic success will vary by form of NCC, but be based upon improvement followed by radiologic stability or slo... | Throughout the course of the study.
To enumerate complications associated with NCC or treatment type for each form of NCC | Throughout the course of the study.
To characterize and correlate the clinical features, radiographic findings, antigen presence and levels, and antibody responses for NCC with perilesional edema | Throughout the course of the study.
To assess diagnostic parameters of serology and antigen detection assays in North American patients | Throughout the course of the study.
To correlate antigen levels in serum and CSF with burden of disease and recurrence of disease in subjects with NCC | Throughout the course of the study.
To characterize cognitive function at baseline, 6, 12, and 24 months as assessed by the Montreal Cognitive Assessment (MOCA) test | Throughout the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Mahanty, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Nash TE, Garcia HH. Diagnosis and treatment of neurocysticercosis. Nat Rev Neurol. 2011 Sep 13;7(10):584-94. doi: 10.1038/nrneurol.2011.135. PMID 21912406
- [Background] Nash T. Edema surrounding calcified intracranial cysticerci: clinical manifestations, natural history, and treatment. Pathog Glob Health. 2012 Sep;106(5):275-9. doi: 10.1179/2047773212Y.0000000026. PMID 23265551
- [Background] Fleury A, Carrillo-Mezo R, Flisser A, Sciutto E, Corona T. Subarachnoid basal neurocysticercosis: a focus on the most severe form of the disease. Expert Rev Anti Infect Ther. 2011 Jan;9(1):123-33. doi: 10.1586/eri.10.150. PMID 21171883